CLINICAL TRIAL: NCT05016297
Title: A Multi-center, Prospective, Open-label, Randomized Study to Explore Efficacy and Safety of Baricitinib in Active Primary Sjogren's Syndrome Patients
Brief Title: Efficacy and Safety of Baricitinib in Sjogren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PekingUMCH-HS-3023D
Record Dates: First submitted 2021-06-26; First posted 2021-08-23 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Sjogren's Syndrome
Keywords: Sjogren's Syndrome; JAK inhibitor; baricitinib; ESSDAI
MeSH Terms: conditions — Sjogren's Syndrome | interventions — baricitinib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- baricitinib 4mg per day + HCQ 200mg twice a day (Experimental): On the basis of the HCQ treatment before, patients in this group will be added on baricitinib 4mg once a day.
  Interventions: Drug: Baricitinib; Drug: Hydroxychloroquine
- HCQ 200mg twice a day (Active Comparator): Patients in this group will be given HCQ 200mg twice a day for 12 weeks. Patients who has no response to HCQ treatment alone at week 12 will be switched to baricitinib + HCQ group and added on baricitinib 4mg per day until the end of the study (week 24).
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Baricitinib — baricitinib 4mg per day
  Arms: baricitinib 4mg per day + HCQ 200mg twice a day
Drug: Hydroxychloroquine — Hydroxychloroquine 200mg twice a day

SUMMARY:
The investigators had observed that baricitinib was effective and safe in active pSS patients in a pilot study. So the investigators plan to conduct a multi-center, prospective, open-label, randomized study to compare the efficacy of baricitinib + hydroxychloroquine (HCQ) with HCQ alone in active pSS patients. The participants will be randomized (1:2) to receive HCQ (200mg twice a day) or baricitinib (4mg per day) + HCQ (200mg twice a day) until week 24. The primary endpoint is the ESSDAI and ESSPRI response (define as an improvement of ESSDAI at least three points, and ESSPRI at least one point or 15%) at 12 weeks. According to an expected response rate of 70% in baricitinib + HCQ group and 30% in HCQ group, the investigators will involve approximately 87 participants (29:58) with 20% drop out rate. The investigators will switch HCQ to baricitinib + HCQ if the participants has no response at 12 weeks. The investigators hypothesized that baricitinib was effective and safe in active pSS patients.

DETAILED DESCRIPTION:
All participants will be divided into HCQ group or HCQ + baricitinib group randomly. On the basis of the HCQ treatment before, the participants in the latter group will be given baricitinib 4mg once a day.

The participants will come to visit at week 0, 4, 8, 12, 16, 20 and 24. The final evaluation will be at week 24. The participants who has no response to HCQ treatment alone at week 12 will be switched to baricitinib + HCQ group and treated with baricitinib 4mg per day until the end of the study (week 24).

Baseline information included demographics, SS duration, clinical manifestations, laboratory parameters, current medications, and disease activity. Laboratory tests, including complete blood counts, urinalysis, liver and renal function tests, ESR, and IgG test were performed at each visit. Disease activity was assessed using the ESSDAI, EULAR primary SS patient reported index (ESSPRI), and physician global assessment (PGA) scores.

ELIGIBILITY:
Inclusion Criteria:

1. Must read and understand the informed consent approved by the institutional review board (IRB)/ethics review board (ERB) governing the site and provide written informed consent.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Ability to take oral medication and be willing to adhere to the study intervention regimen.
4. Male or female, aged between 18-75 years.
5. Fulfill the 2016 ACR/EULAR classification criteria for primary Sjogren's Syndrome.
6. With moderate activity (ESSDAI≥5) at the screening visit.
7. Nonpregnant, nonbreastfeeding female patient
8. Males with potential for reproduction must agree to practice effective birth control methods described above too.

Exclusion Criteria:

1. Have received any of the following medications:

   1. Biologic treatments for immunologic disease such as etanercept, infliximab, certolizumab, adalimumab, golimumab, tocilizumab, abatacept, ustekinumab, ixekizumab, secukinumab, or anakinra within 4 weeks of screening.
   2. Cyclophosphamide (or any other cytotoxic agent), belimumab, or anifrolumab (or another anti-IFN therapy) within 12 weeks of screening.
   3. Rituximab, any other B cell depleting therapies, or intravenous immunoglobulin (IVIg), or pulse methylprednisolone within 24 weeks of screening.
2. Have received treatment with glucocorticoids, methotrexate, azathioprine, mycophenolate mofetil, cyclosporine, tacrolimus within 4 weeks at the time of screening.
3. Have received plasmapheresis within 12 weeks of screening.
4. Have received hemodialysis, peritoneal dialysis, or intestinal dialysis.
5. History of chronic liver disease or elevated LFTs:

   * ALT or AST > 2 x upper limit of normal at screening
   * Serum total bilirubin ≥ 1.5 x upper limit of normal at screening
6. eGFR <40 mL/min/1.73 m2 (Bedside Schwartz formula 2009).
7. Protein to creatinine ratio of more than 1mg/dL repeated and confirmed three times or confirmed with 24 hours urine protein of more than 1000 mg.
8. WBC<2000/microliter or ANC<1,000/microliter, Hgb<9.0 g/dL or platelets <100,000/microliter or absolute lymphocyte count< 500/microliter.
9. Have screening laboratory test values, including thyroid-stimulating hormone (TSH), outside the reference range for the population that, in the opinion of the investigator, pose an unacceptable risk for the patient's participation in the study. Patients who are receiving thyroxine as replacement therapy may participate in the study, provided stable therapy has been administered for ≥12 weeks and TSH is within the laboratory's reference range. Patients who have TSH marginally outside the laboratory's normal reference range and are receiving stable thyroxine replacement therapy may participate if the treating physician has documented that the thyroxine replacement therapy is adequate for the patient.
10. Pregnant or lactating women. Women of childbearing potential are required to have a negative pregnancy test at screening.
11. Have had any major surgery within 8 weeks prior to screening or will require major surgery during the study that, in the opinion of the investigator would pose an unacceptable risk to the patient.
12. Have experienced any of the following within 12 weeks of screening: VTE (DVT/pulmonary embolism [PE]), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
13. Have a history of recurrent (≥ 2) VTE (DVT/PE).
14. Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data.
15. Have a history of lymphoproliferative disease; have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for <5 years prior to randomization.

    The following may be exempted:
    1. Patients with cervical carcinoma in situ that has been resected with no evidence of recurrence or metastatic disease for at least 3 years may participate in the study.
    2. Patients with basal cell or squamous epithelial skin cancers that have been completely resected with no evidence of recurrence for at least 3 years may participate in the study.
16. Have a current or recent (<4 weeks prior to randomization) clinically serious viral, bacterial, fungal, or parasitic infection or any other active or recent infection that in the opinion of the investigator, would pose an unacceptable risk to the patient if participating in the study.

    Note: For example, a recent viral upper respiratory tract infection or uncomplicated urinary tract infection need not be considered clinically serious.
17. Have symptomatic herpes simplex at the time of randomization.
18. Have had symptomatic herpes zoster infection within 12 weeks prior to randomization.
19. Have a history of disseminated/complicated herpes zoster (for example, ophthalmic zoster or CNS involvement).
20. Have a positive test for hepatitis B virus (HBV) defined as:

    1. positive for hepatitis B surface antigen (HBsAg), or
    2. positive for hepatitis B core antibody (HBcAb) and positive for hepatitis B virus deoxyribonucleic acid (HBV DNA) Note: Patients who are HBcAb-positive and HBV DNA-negative may be enrolled in the study but will require additional HBV DNA monitoring during the study.
21. Have hepatitis C virus (HCV) infection (hepatitis C antibody-positive and HCV ribonucleic acid [RNA]-positive).

    Note: Patients who have documented anti-HCV treatment for a past HCV infection AND are HCV RNA-negative may be enrolled in the study.
22. Have evidence of HIV infection and/or positive HIV antibodies.
23. Have had household contact with a person with active TB and did not receive appropriate and documented prophylaxis for TB.
24. Have evidence of active TB or latent TB

    1. Have evidence of active TB, defined in this study as the following:

       * Positive purified protein derivative (PPD) test (≥5 mm induration between approximately 2 and 3 days after application, regardless of vaccination history), medical history, clinical features, and abnormal chest x-ray at screening.
       * QuantiFERON®-TB Gold test or T-SPOT®.TB test (as available and if compliant with local TB guidelines) may be used instead of the PPD test. Patients are excluded from the study if the test is not negative and there is clinical evidence of active TB.

       Exception: patients with a history of active TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, have no clinical features of active TB, and have a screening chest x-ray with no evidence of active TB may be enrolled if other entry criteria met. Such patients would not be required to undergo the protocol-specific TB testing for PPD, QuantiFERON®-TB Gold test, or T-SPOT®.TB test but must have a chest x-ray at screening (i.e., chest imaging performed within the past 6 months will not be accepted).
    2. Have evidence of untreated/inadequately or inappropriately treated latent TB, defined in this study as the following:

       * Positive PPD test, no clinical features consistent with active TB, and a chest x-ray with no evidence of active TB at screening; or
       * If the PPD test is positive and the patient has no medical history or chest x-ray findings consistent with active TB, the patient may have a QuantiFERON®-TB Gold test or T-SPOT®.TB test (as available and if compliant with local TB guidelines). If the test results are not negative, the patient will be considered to have latent TB (for purposes of this study); or
       * QuantiFERON®-TB Gold test or T- SPOT®.TB test (as available and if compliant with local TB guidelines) may be used instead of the PPD test. If the test results are positive, the patient will be considered to have latent TB. If the test is not negative, the test may be repeated once within approximately 2 weeks of the initial value. If the repeat test results are again not negative, the patient will be considered to have latent TB (for purposes of this study).

    Exception: Patients who have evidence of latent TB may be enrolled if he or she completes at least 4 weeks of appropriate treatment prior to randomization and agrees to complete the remainder of treatment while in the trial.

    Exception: Patients with a history of latent TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, have no clinical features of active TB, and have a screening chest x-ray with no evidence of active TB may be enrolled if other entry criteria met. Such patients would not be required to undergo the protocol-specific TB testing for PPD, QuantiFERON®-TB Gold test, or T-SPOT®.TB test but must have a chest x-ray at screening (i.e., chest imaging performed within the past 6 months will not be accepted).
25. Have been exposed to a live vaccine within 12 weeks of randomization or are expected to need/receive a live vaccine during the course of the study (with the exception of herpes zoster vaccination).

    Note: All patients who have not previously received the herpes zoster vaccine by screening will be encouraged (per local guidelines) to do so prior to randomization; vaccination with live herpes zoster vaccine must occur >4 weeks prior to randomization and start of investigational product. Patients will not be randomized if they were exposed to a live herpes zoster vaccination within 4 weeks of planned randomization. Investigators should review the vaccination status of their patients and follow the local guidelines for vaccination of patients ≥18 years of age with non-live vaccines intended to prevent infectious disease prior to entering patients into the study.
26. Are currently enrolled in or have discontinued within 4 weeks of screening from any other clinical trial involving an investigational product or nonapproved use of a drug or device or any other type of medical research judged not to be scientifically or medically compatible with this study.
27. Participants with active renal or central nervous system disease.
28. Significant impairment of major organ function (lung, heart, liver, kidney) or any condition that, in the opinion of the Investigator, would jeopardize the participant's safety following exposure to the study drug.
29. Psychiatric illness or history of medical non-compliance that the study team feels will make the patient unlikely to complete the study.
30. Known allergic reactions to baricitinib or its components.
31. Are largely or wholly incapacitated permitting little or no self-care, such as being bedridden or confined to wheelchair.
32. In the opinion of the investigator, are at an unacceptable risk for participating in the study.
33. Have donated more than a single unit of blood within 4 weeks prior to screening or intend to donate blood during the course of the study.
34. Have a history of intravenous drug abuse, other illicit drug abuse, or chronic alcohol abuse within the 2 years prior to screening or are concurrently using, or expected to use during the study, illicit drugs (including marijuana).
35. Are unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow study restrictions/procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Rate of MCII of ESSDAI | 12 weeks
  The rate of ESSDAI response, or clinically important improvement (MCII) of ESSDAI, which was defined as an improvement of ESSDAI at least three points.

SECONDARY OUTCOMES:
Rate of MCII of ESSDAI | 24 weeks
  The rate of ESSDAI response, or clinically important improvement (MCII) of ESSDAI, which was defined as an improvement of ESSDAI at least three points.
Rate MCII of ESSPRI | 12 and 24 weeks
  The rate of ESSPRI response, or clinically important improvement (MCII) of ESSPRI, which was defined as an improvement of ESSPRI at least one point or 15%.
Change of PGA score | 12 and 24 weeks
  The change from baseline in Physician's Global Assessment (PGA) of disease activity (the minimum value is 0 and maximum value is 3, and higher scores mean a worse outcome) at 12 and 24 weeks.
Change of C-reactive protein (CRP) level | 12 and 24 weeks
  The change from baseline in C-reactive protein (CRP) (mg/L) level at 12 and 24 weeks.
Change of erythrocyte sedimentation rate (ESR) level | 12 and 24 weeks
  The change from baseline in erythrocyte sedimentation rate (ESR) (mm/h) level at 12 and 24 weeks.
Change of immunoglobulin G level | 12 and 24 weeks
  The change from baseline in immunoglobulin G (g/L) level at 12 and 24 weeks.
Change of rheumatoid factor (RF) level | 12 and 24 weeks
  The change from baseline in rheumatoid factor (RF) (IU/ml) level at 12 and 24 weeks.
Change of salivary glands function | 12 and 24 weeks
  The change from baseline in the salivary flow rates (ml/min) at 12 and 24 weeks.
Change of lacrimal glands function | 12 and 24 weeks
  The change from baseline in the Schirmer's test (mm) at 12 and 24 weeks.
Change of focus score on labial salivary gland biopsy | 24 weeks
  The change from baseline in the focus score on labial salivary gland biopsy (the minimum value is 1 and maximum value is 12, and higher scores mean a worse outcome) at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Leng, Dr., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 5 years after article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to lengxm@gmail.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Bai W, Yang F, Xu H, Wei W, Li H, Zhang L, Zhao Y, Shi X, Zhang Y, Zeng X, Leng X. A multi-center, open-label, randomized study to explore efficacy and safety of baricitinib in active primary Sjogren's syndrome patients. Trials. 2023 Feb 15;24(1):112. doi: 10.1186/s13063-023-07087-5. PMID 36793118